CLINICAL TRIAL: NCT01499511
Title: Anglo-Scandinavian Cardiac Outcomes Trial: Post Trial Follow-Up Study
Acronym: ASCOT-10
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CRO1667; 2010-023875-24 (EudraCT Number)
Record Dates: First submitted 2011-02-07; First posted 2011-12-26 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Hypertension; Diabetes; Death From Cardiovascular Disease; Myocardial Infarction; Stroke
Keywords: Hypertension; Mortality; Morbidity; Coronary Heart Disease; Stroke; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Myocardial Infarction; Stroke; Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma to be stored for future measurement of biochemical markers of cardiovascular disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASCOT participants amlodipine: It is follow up group from the ASCOT study, after treatment with amlodipine for 5.5 years. No treatment only follow up.
- ASCOT participants atenolol: It is follow up group from the ASCOT study, after treatment with atenolol for 5.5 years. No treatment only follow up.

SUMMARY:
ASCOT-10 is a follow-up study of surviving participants in the United Kingdom (UK)arm of the Anglo-Scandinavian Cardiac Outcomes Trial (ASCOT) which was conducted between 2000 and 2005.ASCOT's results showed substantial cardiovascular benefit from: 1) the use of a cholesterol lowering drug (atorvastatin) compared to placebo, and 2) the use of a blood-pressure lowering strategy based on amlodipine when compared to a strategy based on atenolol. ASCOT-10 will test the hypothesis that the ASCOT subjects who originally received Atorvastatin and those who received amlodipine based treatment will continue to show a cardiovascular benefit relative to those who did not, even though all the subjects have had access to optimal treatment in the interim.

DETAILED DESCRIPTION:
Study investigators will have access to information about ASCOT patients from their study centre who have died since the end of the ASCOT study in 2005. Of the 8580 ASCOT patients from the United Kingdom, 7300 were flagged with The Information Centre for Health and Social Care at the end of the trial in 2005.This flagging process was re-activated in 2010 so that all deaths and incident cancers relating to these patients are now sent every three months to the ASCOT-10 co-ordinating centre. These results are identified by the ASCOT study number, with all personal data removed. These deceased patient numbers will be communicated to the participating sites so that the trial centre staff will not contact their families.

An attempt will be made to contact all remaining patients from the participating UK ASCOT sites.

Initial contact will be made via the general practitioner (GP) surgery. If the GP can provide up-to-date contact details and feels that it is appropriate to contact the patient, patients will then be sent an introductory letter, a patient information sheet, a consent form and a health questionnaire.

They will be asked to complete a 'tick-box' form given the following options:

1. Willing to complete health questionnaire.
2. Willing for information about health to be given by GP or next of kin.
3. Willing to give information by telephone only.
4. Willing to attend study clinic for a single visit.
5. Not willing to take part.

They will be asked to complete this form, sign, date and return in a pre-paid envelope to their trial centre. This form will be used as the consent form for the questionnaire part of the study.

They will also be asked to complete a simple health questionnaire. This will collect information on any health problems experienced since the end of the ASCOT trial (in particular about heart attacks and strokes/mini-strokes), as well as information on any hospital admissions during this period and current medication. In addition, information about current weight, exercise, alcohol consumption, smoking and general quality of life will be collected. Patients will be asked to return their completed questionnaire, along with their consent/reply form, to their local trial centre.

If the study team have not received a response within four weeks, a further reminder letter will be sent. If no response has been obtained after a further four weeks, a final attempt will be made to contact the patient by letter or telephone call.

10% of the study population from each trial centre, who will be chosen at random, will be invited to attend their trial centre for a single clinic visit. Further informed consent following discussion with member(s) of the study team will be obtained. During the clinic visit the questionnaire will be reviewed and several further measurements will be taken as follows:

* Blood pressure
* Weight
* Pulse wave analysis. (This is a simple, non-invasive test, very much like a blood pressure measurement, that gives us further information on the function of the heart and arteries)
* Blood for creatinine and estimated glomerular filtration rate(eGFR)(tests of kidney function), electrolytes (sodium and potassium), fasting lipids (cholesterol), fasting glucose, glycated haemoglobin (a further test for diabetes) An additional blood test will be taken and plasma stored for the later analysis of chemicals in the blood which might predict cardiovascular risk. Precise details of this further testing are not currently available. However, the plasma will be stored securely and no identifiable data will be present on the samples (i.e. they will be stored anonymously, identified only by the subject's study number).

Every effort will be taken to contact patients who have moved since the ASCOT study closed and for whom no contact details are available. This may be done by health service tracking services, where available, or via Primary Care Trusts (PCTs).

ELIGIBILITY:
Inclusion Criteria:

* Surviving ASCOT participants from the participating UK sites

Exclusion Criteria:

* None

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who participated in the Anglo-Scandinavian Cardiac Outcomes Trial in the UK
Sampling Method: Non-Probability Sample
Enrollment: 1718 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2016-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Mackay, MBBS PhD MRCP, Study Director — Imperial College Healthcare NHS Trust; Peter S Sever, MBChB FRCP PhD, Principal Investigator — Imperial College London; Simon M Thom, MBBS MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- International Centre for Circulatory Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahlof B, Sever PS, Poulter NR, Wedel H, Beevers DG, Caulfield M, Collins R, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J; ASCOT Investigators. Prevention of cardiovascular events with an antihypertensive regimen of amlodipine adding perindopril as required versus atenolol adding bendroflumethiazide as required, in the Anglo-Scandinavian Cardiac Outcomes Trial-Blood Pressure Lowering Arm (ASCOT-BPLA): a multicentre randomised controlled trial. Lancet. 2005 Sep 10-16;366(9489):895-906. doi: 10.1016/S0140-6736(05)67185-1. PMID 16154016

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
Started | 885 | 833
Completed | 884 | 833
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients recruited into long term follow up
Groups:
- Total: Total of all reporting groups
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol | Total
Number analyzed (Participants) | 885 | 833 | 1718
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 88 | 173
  >=65 years | 800 | 745 | 1545
Age, Continuous [Median (Full Range); unit: years] | 75 [54 to 93] | 74.5 [52 to 91] | 74.8 [52 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 739 | 720 | 1459
  Male | 146 | 113 | 259
Region of Enrollment [Number; unit: participants]
  United Kingdom | 885 | 833 | 1718

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have Died From Cardiovascular Disease Since the End of the ASCOT Study
Description: Number of participants who have died from cardiovascular disease since the end of the Anglo-Scandinavian Cardiac Outcomes Trial-Blood Pressure Lowering Armstudy
Time Frame: 16 years
Population: Data not collected
Groups:
- ASCOT Participants: Participants from the ASCOT study recruited to the participating ASCOT study centres in the United Kingdom.
Arm/Group | ASCOT Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Non Fatal Myocardial Infarction
Description: Morbidity of non fatal myocardial infarction after 16 years in patients recruited into the Anglo-Scandinavian Outcomes trial with two groups
Time Frame: 16 years
Population: 13 participants had missing data
Measure: Count of Participants; unit: Participants
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
Number analyzed (Participants) | 877 | 828
Participants | 35 | 37
Statistical Analysis 1: Comparison: ASCOT Participants Amlodipine vs ASCOT Participants Atenolol; Test type: Superiority; p = 0.624, ANOVA

3. Primary Outcome: Number of Participants With Non Fatal Stroke/TIA (Transient Ischaemic Attack)
Description: Non fatal stroke and TIA (Transient Ischaemic Attack) morbidity after 16 years in patients recruited into the Anglo-Scandinavian Outcomes trial
Time Frame: 16 years
Population: 18 participants had missing data
Measure: Count of Participants; unit: Participants
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
Number analyzed (Participants) | 877 | 823
Participants | 29 | 52
Statistical Analysis 1: Comparison: ASCOT Participants Amlodipine vs ASCOT Participants Atenolol; Test type: Superiority; p = 0.004, ANOVA

4. Secondary Outcome: Number of Participants Who Have Developed Diabetes Since the End of the ASCOT Trial
Description: Diabetes morbidity after 16 years in patients recruited into the Anglo-Scandinavian Outcomes trial
Time Frame: 16 years
Population: 22 participants had missing data
Measure: Count of Participants; unit: Participants
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
Number analyzed (Participants) | 871 | 825
Participants | 322 | 325
Statistical Analysis 1: Comparison: ASCOT Participants Amlodipine vs ASCOT Participants Atenolol; Test type: Superiority; p = 0.304, ANOVA

5. Secondary Outcome: Number of Participants Who Have Undergone Coronary/Peripheral Re-vascularisation Procedures Since the End of the ASCOT Trial
Description: Number of participants who have undergone coronary/peripheral re-vascularisation procedures since the end of the ASCOT trial, follow up
Time Frame: 16 years
Population: 24 participants had missing data
Measure: Count of Participants; unit: Participants
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
Number analyzed (Participants) | 872 | 822
Participants | 39 | 33
Statistical Analysis 1: Comparison: ASCOT Participants Amlodipine vs ASCOT Participants Atenolol; Test type: Superiority; p = 0.641, ANOVA

6. Secondary Outcome: Number of Participants Who Have Required Renal Replacement Therapy (Dialysis or Kidney Transplant) Since the End of the ASCOT Trial
Description: Number of participants who have required renal replacement therapy (dialysis or kidney transplant) since the end of the ASCOT trial, follow up
Time Frame: 16 years
Population: 18 participants had missing data
Measure: Count of Participants; unit: Participants
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
Number analyzed (Participants) | 874 | 826
Participants | 10 | 9
Statistical Analysis 1: Comparison: ASCOT Participants Amlodipine vs ASCOT Participants Atenolol; Test type: Superiority; p = 0.915, ANOVA

7. Secondary Outcome: Number of Participants Who Have Experienced a Transient Ischaemic Attack (TIA) Since the End of the ASCOT Trial
Time Frame: 16 years
Population: Combined together with 3. primary outcome, it was not possible to differentiate between data collected for TIAs and Non fatal stroke
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 years
Groups:
- ASCOT Participants Amlodipine: Follow up study for amlodipine, no intervention.
- ASCOT Participants Atenolol: Follow up study for atenolol, no intervention.
Arm/Group | ASCOT Participants Amlodipine | ASCOT Participants Atenolol
All-Cause Mortality (participants affected / at risk) | 1/885 | 0/833
Serious Adverse Events (participants affected / at risk) | 2/885 | 0/833
Other Adverse Events (participants affected / at risk) | 4/885 | 1/833
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASCOT Participants Amlodipine (N=885) | ASCOT Participants Atenolol (N=833)
Injuries (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — after fall from bicycle
Ischaemic stroke (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASCOT Participants Amlodipine (N=885) | ASCOT Participants Atenolol (N=833)
Collapse (Nervous system disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stomach cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
High blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Alcohol dependence withdrawal (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes